CLINICAL TRIAL: NCT03443414
Title: Phase IIb, Randomized, Double Blind, Placebo Controlled, Dose Ranging Study to Assess the Effect of RPL554 in Patients With Moderate to Severe COPD.
Brief Title: Dose Ranging Study of RPL554 in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RPL554-CO-203
Record Dates: First submitted 2018-02-07; First posted 2018-02-23 (Actual); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: COPD
Keywords: COPD, bronchodilation, FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The nebuliser cup will be obscured to prevent the Investigator or outcomes assessor so the contents are not visible to the Investigator our outcomes assessor. The visual appearance of the study medication will not be discussed with the subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 0.75 mg RPL554 (Experimental)
  Interventions: Drug: RPL554 suspension
- 1.5 mg RPL554 (Experimental)
  Interventions: Drug: RPL554 suspension
- 3 mg RPL554 (Experimental)
  Interventions: Drug: RPL554 suspension
- 6 mg RPL554 (Experimental)
  Interventions: Drug: RPL554 suspension
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPL554 suspension — A dual PDE3/PDE 4 inhibitor
  Arms: 0.75 mg RPL554; 1.5 mg RPL554; 3 mg RPL554; 6 mg RPL554
Drug: Placebo — Placebo solution
  Arms: Placebo

SUMMARY:
The study investigates the effect of 4 weeks of twice daily treatment of four different doses of RPL554 (a phosphodiesterase [PDE]3/4 inhibitor) or placebo in patients with moderate to severe chronic obstructive pulmonary disease (COPD). Patients will be equally allocated to one of the five treatment options.

DETAILED DESCRIPTION:
RPL554 is a dual inhibitor of PDE3 and PDE4 which are known to have a role in modulating the inflammatory airway response in respiratory diseases, including COPD. PDE3 inhibitors act as bronchodilators whilst PDE4 inhibitors have anti-inflammatory properties and there is also evidence to suggest that combined inhibition of PDE3 and PDE4 can have additive or synergistic anti-inflammatory and bronchodilator effects. PDE4 inhibitors (administered orally) have, however been associated with unfavorable gastrointestinal side effects such as nausea, emesis, diarrhea, abdominal pain, loss of appetite and weight loss. Dual PDE3/PDE4 inhibitors (administered by inhalation) have exhibited both bronchodilator and anti-inflammatory actions, with a more favorable side effect profile. It is plausible that increased efficacy with reduced side effects may be achievable with administration of a dual PDE3/4 inhibitor by the inhaled route compared to orally administered PDE3 or PDE4 inhibitors.

The purpose of this study is to investigate the dose response of RPL554 in patients with COPD over 4 weeks. This length of time should allow for study of the bronchodilator response, measured predominantly by the peak forced expiratory volume in one second (FEV1), and the anti-inflammatory response, as measured predominantly by trough FEV1.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Male or female aged 40 to 75 years
* Meeting specified contraception requirements
* 12-lead electrocardiogram with heart rate 50-90 beats per minute, QT interval corrected using Fridericia's formula (QTcF) ≤450 msec (males) or ≤470 msec (females), QRS interval ≤120 msec, PR interval ≤200 msec and no clinically significant abnormalities
* Capable of complying with all study restrictions and procedures, including ability to use the study nebulizer correctly.
* Body mass index (BMI) 18 to 35 kg/m2 and minimum weight 45 kg.
* COPD diagnosis with symptoms compatible with COPD for at least 1 year
* Clinically stable COPD in the previous 4 weeks
* Ability to perform acceptable and reproducible spirometry.
* Post-bronchodilator spirometry at screening must demonstrate FEV1/forced vital capacity (FVC) ratio of ≤0.70 and FEV1 must be ≥40 % to ≤80% of predicted normal
* Chest X-ray (posterior-anterior) at screening, or chest X-ray, magnetic resonance imaging (MRI) or computed tomography (CT) scan in the last 12 months, showing no abnormalities which are both clinically significant and unrelated to COPD.
* Meet the concomitant medication restrictions and be expected to do so for the rest of the study.
* Current and former smokers with a smoking history of ≥10 pack years.
* Capable of withdrawing long acting bronchodilators until the end of the treatment period, and short acting bronchodilators for 8 hours prior to administration of study medication.

Exclusion Criteria:

* A history of life-threatening COPD including Intensive Care Unit admission and requiring intubation.
* COPD exacerbation requiring oral steroids in the previous 3 months
* A history of one or more hospitalizations for COPD in the previous 6 months
* Lower respiratory tract infection treated with antibiotics in the previous 3 months
* Evidence of cor pulmonale or clinically significant pulmonary hypertension.
* Patients with a current diagnosis of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, sleep apnea, known alpha-1 antitrypsin deficiency or other active pulmonary diseases.
* Previous lung resection or lung reduction surgery.
* Oral therapies for COPD (e.g. oral steroids, theophylline, and roflumilast) in the previous 3 months and throughout the study.
* Pulmonary rehabilitation, unless such treatment has been stable from 4 weeks prior to Visit 1) and remains stable during the trial.
* A history of, or reason to believe a subject has, drug or alcohol abuse in the previous 3 years.
* Received an experimental drug within 30 days or five half-lives of the first dose
* Prior exposure to RPL554.
* Women who are pregnant or breast-feeding.
* Patients with a history of current uncontrolled disease that the Investigator believes are clinically significant.
* myocardial infarction in the previous 6 month; congestive heart failure, a history of unstable or uncontrolled hypertension, or has been diagnosed with hypertension in last 3 months.
* Use of oral beta blockers.
* Major surgery (requiring general anesthesia) in the previous 6 weeks, lack of full recovery from surgery at screening, or planned surgery through the end of the study.
* History of malignancy of any organ system within 5 years, with the exception of localized skin cancers (basal or squamous cell).
* Clinically significant abnormal values for safety laboratory tests
* Significant non-compliance in previous investigational studies or with prescribed medications.
* Requirement for oxygen therapy, even on an occasional basis.
* Known hypersensitivity to RPL554 or its excipients/components.
* Abnormal clinically significant 12 lead Holter findings,
* Any other reason that the Investigator considers makes the subject unsuitable to participate.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Singh, Principal Investigator — Medicines Evaluation Unit (MEU)
Locations (49):
- Bulgaria (8):
  - Clinic for pneumonology, Pleven
  - SHATPPD-Ruse EOOD, Rousse
  - Fifth MHAT - Sofia EAD, Sofia
  - MHAT 'Lyulin', EAD, Sofia
  - NMTH Tsar Boris III, Sofia
  - UMHAT 'Alexandrovska' EAD, Sofia
  - UMHAT 'Sveta Anna' AD, Sofia
  - Medical Center Nov, Stara Zagora
- Czechia (2):
  - MediTrial s.r.o., Jindřichův Hradec
  - Plicni stredisko Teplice, Teplice
- Germany (17):
  - Aerzte fuer Lungen- und, Berlin
  - Charite Campus Mitte, Berlin
  - emovis GmbH, Berlin
  - Studienpraxis Berlin, Berlin
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Praxis Dr. Keller, Frankfurt
  - Inamed GmbH, Gauting
  - PRI Pulmonary Research, Großhansdorf
  - Hamburger Institut fuer, Hamburg
  - Gemeinschaftspraxis Dres, Koblenz
  - POIS Leipzig GbR, Leipzig
  - SALVUS UG Centre for Clinial Trials, Leipzig
  - KLB Gesundheitsforschung, Lübeck
  - Pneumologie Odeonsplatz, Munich
  - Pneumologische Praxis Pasing, München
  - Ballenberger Freytag Wenisch, Neu-Isenburg
  - Dr. Christian Schlenska, Peine
- Poland (14):
  - CERMED, Bialystok
  - Indywidualna Specjalistyczna, Bialystok
  - KLIMED Marek Klimkiewicz, Bychawa
  - Silmedic sp. z o.o., Katowice
  - Grazyna Pulka Specjalistyczny, Krakow
  - Malopolskie Centrum Alergologii, Krakow
  - Centrum Terapii Wspólczesnej, Lodz
  - Uniwersytecki Szpital Klin, Lodz
  - NZOZ Alergo-MEDSpecjalistyczna, Poznan
  - ETG Network Sp z o o, Skierniewice
  - Centrum Medyczne Pratia, Warsaw
  - Mazowieckie Centrum Medyczne, Warsaw
  - Centrum Badan Klinicznych, Wroclaw
  - Specjalistyczna Opieka, Wroclaw
- Romania (7):
  - S.C Angisan S.R.L, Bragadiru
  - S.C Clinica Pneumomedica S.R.L, Brasov
  - Fundatia Dr. Victor Babes, Bucharest
  - Spitalul Clinic de Urgenta, Bucharest
  - Spitalul Cl. Pneumoftiziologie, Cluj-Napoca
  - Spitalul CldePneumoftiziologie, Constanța
  - Spitalul CldePneumoftiziologie, Iași
- Medicines Evaluation Unit, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 405 adult patients with moderate to severe chronic obstructive pulmonary disease (COPD) were randomized into this double-blind, multicenter study, and 403 received study medication. Patients were recruited to 47 study centers in Bulgaria, Czech Republic, Germany, Poland, Romania and the United Kingdom.
Pre-assignment Details: Patients with a clinical diagnosis of COPD as defined by the American Thoracic Society/European Respiratory Society guidelines with symptoms compatible with COPD for at least 1 year prior to screening, and with clinically stable symptoms in the 4 weeks prior to screening and randomization were screened for inclusion.
Groups:
- RPL554 0.75 mg: Patients were randomized to receive 0.75 milligrams (mg) RPL554 administered by jet nebulizer twice daily (morning and evening) for 4 weeks.
- RPL554 1.5 mg: Patients were randomized to receive 1.5 mg RPL554 administered by jet nebulizer twice daily (morning and evening) for 4 weeks.
- RPL554 3.0 mg: Patients were randomized to receive 3.0 mg RPL554 administered by jet nebulizer twice daily (morning and evening) for 4 weeks.
- RPL554 6.0 mg: Patients were randomized to receive 6.0 mg RPL554 administered by jet nebulizer twice daily (morning and evening) for 4 weeks.
- Placebo: Patients were randomized to receive placebo administered by jet nebulizer twice daily (morning and evening) for 4 weeks.
Period: Overall Study
Arm/Group | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | RPL554 6.0 mg | Placebo
Started | 82 | 81 | 82 | 80 | 80
Received Treatment | 81 | 81 | 82 | 80 | 79
Completed | 71 | 78 | 76 | 75 | 75
Not Completed | 11 | 3 | 6 | 5 | 5
Not completed — Adverse Event | 6 | 0 | 4 | 2 | 3
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 2 | 1
Not completed — Death | 0 | 1 | 0 | 1 | 0
Not completed — Reason not specified | 2 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline population consists of all randomized patients.
Groups:
- RPL554 0.75 mg: Patients were randomized to receive 0.75 mg RPL554 administered by jet nebulizer twice daily (morning and evening) for 4 weeks.
Arm/Group | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | RPL554 6.0 mg | Placebo | Total Title
Number analyzed (Participants) | 82 | 81 | 82 | 80 | 80 | 405
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (7.05) | 63.4 (6.40) | 62.5 (6.51) | 62.9 (6.73) | 63.5 (6.44) | 63.2 (6.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 35 | 37 | 32 | 30 | 160
  Male | 56 | 46 | 45 | 48 | 50 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 82 | 81 | 82 | 80 | 80 | 405
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 82 | 81 | 82 | 80 | 80 | 405
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Peak FEV1 (Over 3 Hours) at Week 4
Description: Spirometry assessments were used to assess pulmonary function including the forced expiratory volume in 1 second (FEV1). Peak FEV1 at Week 4 was defined as the maximum post-dose value among the 30 minutes, 1, 2 and 3 hour assessments collected at Visit 6. Baseline was defined as the FEV1 pre-dose assessment (-15 minutes) collected at Visit 2. A mixed model for repeated measures (MMRM) was used to model the change from baseline FEV1 using baseline FEV1 as a continuous fixed effect, randomized treatment, week and treatment-by-week as categorical fixed effect, and patient as random effect.
  The least squares (LS) mean change from baseline FEV1 to peak FEV1 (as measured over 3 hours) at Week 4 is presented.
Time Frame: Baseline (pre-dose, Visit 2) and Week 4 (Visit 6).
Population: The full analysis set (FAS) consisted of all randomized patients, who received at least 1 dose of investigational product during the study and with at least 1 post-treatment efficacy data assessment. Data is presented for the number of patients with at least 1 on-treatment value who contributed to the model estimate.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | RPL554 6.0 mg | Placebo
Number analyzed (Participants) | 81 | 81 | 82 | 80 | 79
Liters | 0.203 [0.152 to 0.253] | 0.209 [0.160 to 0.258] | 0.257 [0.208 to 0.306] | 0.196 [0.147 to 0.246] | 0.057 [0.007 to 0.106]
Statistical Analysis 1: Comparison: RPL554 6.0 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 6.0 mg - Placebo); Test type: Other — A fixed-sequence testing approach was used, starting with the highest dose versus placebo. If a statistically significant difference was found at the 2-sided alpha level of 5%, the testing proceeded to the next highest dose; p < 0.001, MMRM; LS mean difference = 0.139, 95% CI 2-sided [0.069 to 0.210]
Statistical Analysis 2: Comparison: RPL554 3.0 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 3.0 mg - Placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, MMRM; LS mean difference = 0.200, 95% CI 2-sided [0.131 to 0.270]
Statistical Analysis 3: Comparison: RPL554 1.5 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 1.5 mg - Placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, MMRM; LS mean difference = 0.153, 95% CI 2-sided [0.083 to 0.222]
Statistical Analysis 4: Comparison: RPL554 0.75 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 0.75 mg - Placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, MMRM; LS mean difference = 0.146, 95% CI 2-sided [0.075 to 0.216]

2. Secondary Outcome: Mean Change From Baseline FEV1 to Morning Trough FEV1 at Week 4
Description: Morning trough FEV1 was defined as the last pre-dose value at Visit 6. Baseline was defined as the FEV1 pre-dose assessment (-15 minutes) collected at Visit 2. MMRM was used to model the change from baseline FEV1 using baseline FEV1 as a continuous fixed effect, randomized treatment, week and treatment-by-week as categorical fixed effect, and patient as random effect.
  The LS mean change from baseline FEV1 to morning trough FEV1 at Week 4 is presented.
Time Frame: Baseline (pre-dose, Visit 2) and Week 4 (Visit 6).
Population: The FAS consisted of all randomized patients, who received at least 1 dose of investigational product during the study and with at least 1 post-treatment efficacy data assessment. Data is presented for the number of patients with at least 1 on-treatment value who contributed to the model estimate.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | RPL554 6.0 mg | Placebo
Number analyzed (Participants) | 77 | 80 | 82 | 77 | 78
Liters | 0.007 [-0.038 to 0.053] | -0.019 [-0.063 to 0.025] | 0.040 [-0.003 to 0.084] | -0.026 [-0.071 to 0.018] | -0.028 [-0.072 to 0.016]
Statistical Analysis 1: Comparison: RPL554 6.0 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 6.0 mg - Placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.953, MMRM; LS mean difference = 0.002, 95% CI 2-sided [-0.061 to 0.065]
Statistical Analysis 2: Comparison: RPL554 3.0 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 3.0 mg - Placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.032, MMRM; LS mean difference = 0.068, 95% CI 2-sided [0.006 to 0.130]
Statistical Analysis 3: Comparison: RPL554 1.5 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 1.5 mg - Placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.773, MMRM; LS mean difference = 0.009, 95% CI 2-sided [-0.053 to 0.072]
Statistical Analysis 4: Comparison: RPL554 0.75 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 0.75 mg - Placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.272, MMRM; LS mean difference = 0.035, 95% CI 2-sided [-0.028 to 0.099]

3. Secondary Outcome: Mean Change From Baseline FEV1 to Average FEV1 (Over 12 Hours) at Day 1 and Week 4
Description: Average FEV1 over 12 hours was defined as the area under the curve from 0 to 12 hours post-dose (AUC[0-12]) of the FEV1 values collected during the visit under analysis (Day 1 or Week 4), divided by the length of the time interval of interest (in hours). The AUC was calculated using the trapezoidal rule. Baseline was defined as the FEV1 pre-dose assessment (-15 minutes) collected at Visit 2. MMRM was used to model the change from baseline FEV1 using baseline FEV1 as a continuous fixed effect, randomized treatment, week and treatment-by-week as categorical fixed effect, and patient as random effect.
  The LS mean change from baseline FEV1 to average FEV1 over 12 hours at Day 1 and at Week 4 is presented.
Time Frame: Baseline (pre-dose, Visit 2), up to 12 hours post-dose at Visit 2 (Day 1) and Visit 6 (Week 4).
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | RPL554 6.0 mg | Placebo
Number analyzed (Participants) | 81 | 81 | 82 | 80 | 79
Liters
  Day 1: number analyzed (Participants) | 80 | 81 | 82 | 79 | 78
  Day 1 | 0.088 [0.058 to 0.117] | 0.077 [0.048 to 0.107] | 0.103 [0.074 to 0.132] | 0.095 [0.065 to 0.125] | 0.008 [-0.022 to 0.038]
  Week 4: number analyzed (Participants) | 80 | 81 | 82 | 79 | 78
  Week 4 | 0.039 [-0.007 to 0.085] | 0.052 [0.008 to 0.096] | 0.085 [0.040 to 0.130] | 0.031 [-0.014 to 0.076] | -0.033 [-0.079 to 0.012]
Statistical Analysis 1: Comparison: RPL554 6.0 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 6.0 mg - Placebo) at Day 1; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, MMRM; LS mean difference = 0.087, 95% CI 2-sided [0.045 to 0.129]
Statistical Analysis 2: Comparison: RPL554 3.0 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 3.0 mg - Placebo) at Day 1; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, MMRM; LS mean difference = 0.095, 95% CI 2-sided [0.053 to 0.137]
Statistical Analysis 3: Comparison: RPL554 1.5 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 1.5 mg - Placebo) at Day 1; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.001, MMRM; LS mean difference = 0.070, 95% CI 2-sided [0.028 to 0.112]
Statistical Analysis 4: Comparison: RPL554 0.75 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 0.75 mg - Placebo) at Day 1; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, MMRM; LS mean difference = 0.080, 95% CI 2-sided [0.038 to 0.122]
Statistical Analysis 5: Comparison: RPL554 6.0 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 6.0 mg - Placebo) at Week 4; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.048, MMRM; LS mean difference = 0.065, 95% CI 2-sided [0.001 to 0.129]
Statistical Analysis 6: Comparison: RPL554 3.0 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 3.0 mg - Placebo) at Week 4; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, LS mean difference; LS mean difference = 0.119, 95% CI 2-sided [0.055 to 0.183]
Statistical Analysis 7: Comparison: RPL554 1.5 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 1.5 mg - Placebo) at Week 4; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.008, MMRM; LS mean difference = 0.085, 95% CI 2-sided [0.022 to 0.149]
Statistical Analysis 8: Comparison: RPL554 0.75 mg vs Placebo; Placebo-corrected treatment effect: LS mean difference (RPL554 0.75 mg - Placebo) at Week 4; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.028, MMRM; LS mean difference = 0.072, 95% CI 2-sided [0.008 to 0.137]

4. Secondary Outcome: Mean Change From Baseline in COPD Symptoms Using the Exacerbations of Chronic Pulmonary Disease Tool Patient-Reported Outcome (EXACT-PRO) Scoring at Week 4
Description: Patients completed an electronic diary (e-diary) once daily which used the 14-item EXACT-PRO instrument to assess COPD symptoms. The EXACT-PRO instrument contains 11 respiratory symptom questions that comprise the derivative Evaluating Respiratory Symptoms (E-RS) instrument that was used to measure the effect of treatment with RPL554 on the severity of COPD symptoms overall. The E-RS tool contains 3 subscales to assess breathlessness, cough/sputum and chest symptoms. In addition to the subscale scores, a total score for the E-RS part was obtained. The raw totals for the E-RS score and for each of the subscales were converted to a scale range of 0 to 100 (least symptomatic to most symptomatic). MMRM was used to model the change from baseline using baseline as a continuous fixed effect, randomized treatment, week and treatment-by-week as categorical fixed effect, and patient as random effect. Baseline was the last non-missing assessment taken prior to investigational product start date.
Time Frame: Baseline (pre-dose, Visit 2) and Week 4 (Visit 6).
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | RPL554 6.0 mg | Placebo
Number analyzed (Participants) | 81 | 81 | 82 | 80 | 79
Units on a scale
  E-RS Total Score: number analyzed (Participants) | 71 | 74 | 76 | 74 | 76
  E-RS Total Score | -1.07 [-2.00 to -0.14] | -1.26 [-2.16 to -0.35] | -0.80 [-1.69 to 0.10] | -0.92 [-1.81 to -0.02] | 1.19 [0.30 to 2.08]
  E-RS Breathlessness Score: number analyzed (Participants) | 71 | 74 | 76 | 74 | 76
  E-RS Breathlessness Score | -0.46 [-0.92 to -0.01] | -0.63 [-1.07 to -0.18] | -0.48 [-0.92 to -0.04] | -0.48 [-0.92 to -0.04] | 0.47 [0.03 to 0.90]
  E-RS Cough/Sputum Score: number analyzed (Participants) | 71 | 74 | 76 | 74 | 76
  E-RS Cough/Sputum Score | -0.22 [-0.50 to 0.07] | -0.30 [-0.58 to -0.03] | -0.14 [-0.41 to 0.13] | -0.21 [-0.48 to 0.06] | 0.36 [0.09 to 0.63]
  E-RS Chest Symptoms Score: number analyzed (Participants) | 71 | 74 | 76 | 74 | 76
  E-RS Chest Symptoms Score | -0.39 [-0.70 to -0.08] | -0.32 [-0.62 to -0.02] | -0.19 [-0.48 to 0.11] | -0.22 [-0.52 to 0.07] | 0.35 [0.05 to 0.64]

5. Secondary Outcome: Mean Change From Baseline in Breathlessness as Assessed Using the St George's Respiratory Questionnaire (SGRQ) at Week 4
Description: Patients completed the COPD specific SGRQ (SGRQ-C) consisting of 14 items each weighted from 0 to a possible maximum of 100. Items 1-7 produced the symptoms score, 9-12 the activity score, and items 8, 10, 11, 13 and 14 the impacts score. Each component sub-score was calculated as a percentage of the summed weights of each item out of the sum of the maximum possible weight for that component (range 0-100). The total score was calculated by summing the weights to all positive responses in each component, where a positive item indicated the presence of symptoms, expressed as a percentage (range 0-100). Higher scores indicate a worse outcome. Baseline assessment was pre-dose at Visit 2. MMRM was used to model the change from baseline using baseline as a continuous fixed effect, randomized treatment, week and treatment-by-week as categorical fixed effect, patient as random effect. The LS mean change from baseline in the total, symptoms, activity and impact SGRQ-C scores are presented.
Time Frame: Baseline (pre-dose, Visit 2) and Week 4 (Visit 6).
Population: The FAS consisted of all randomized patients, who received at least 1 dose of investigational product during the study and with at least 1 post-treatment efficacy data assessment. Data is presented for the numbers of patients with at least 1 on-treatment value who contributed to the model estimate.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | RPL554 6.0 mg | Placebo
Number analyzed (Participants) | 81 | 81 | 82 | 80 | 79
Units on a scale
  SGRQ-C Total score: number analyzed (Participants) | 74 | 75 | 71 | 77 | 73
  SGRQ-C Total score | -2.56 [-5.13 to 0.02] | -3.18 [-5.72 to -0.65] | -2.63 [-5.24 to -0.01] | -3.01 [-5.51 to -0.51] | -0.33 [-2.90 to 2.23]
  SGRQ-C Symptoms score: number analyzed (Participants) | 74 | 75 | 71 | 77 | 73
  SGRQ-C Symptoms score | -4.73 [-7.99 to -1.46] | -1.89 [-5.11 to 1.33] | -2.17 [-5.50 to 1.17] | -4.33 [-7.51 to -1.16] | 1.25 [-2.02 to 4.51]
  SGRQ-C Activity score: number analyzed (Participants) | 74 | 75 | 71 | 77 | 73
  SGRQ-C Activity score | -2.19 [-5.30 to 0.91] | -4.28 [-7.34 to -1.23] | -2.70 [-5.85 to 0.46] | -2.75 [-5.76 to 0.27] | -2.16 [-5.25 to 0.94]
  SGRQ-C Impact score: number analyzed (Participants) | 74 | 75 | 71 | 77 | 73
  SGRQ-C Impact score | -1.73 [-4.91 to 1.46] | -2.93 [-6.06 to 0.20] | -2.96 [-6.20 to 0.28] | -2.80 [-5.89 to 0.29] | 0.11 [-3.07 to 3.28]

6. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs)
Description: The number of patients with TEAEs for each the following categories are presented: any TEAE, any drug-related TEAE, any severe TEAE, any serious TEAE, serious drug-related TEAE, any TEAE leading to drug interruption, any TEAE leading to drug discontinuation, and any TEAE leading to death.
  All AEs which started after the first dose of investigational product.or started prior to first dose and worsened, based on the Investigator assessment of severity, on or after first dose were considered to be treatment-emergent.
Time Frame: Up to end of study (approximately 6 weeks)
Population: The safety analysis set consisted of all patients who received at least 1 dose of investigational product during the study.
Measure: Number; unit: Patients
Arm/Group | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | RPL554 6.0 mg | Placebo
Number analyzed (Participants) | 81 | 81 | 82 | 80 | 79
Patients
  Any TEAE | 27 | 36 | 29 | 29 | 31
  Any drug-related TEAE | 8 | 11 | 12 | 8 | 10
  Any severe TEAE | 4 | 1 | 2 | 1 | 2
  Any serious TEAE | 2 | 2 | 1 | 1 | 1
  Any serious drug-related TEAE | 1 | 1 | 0 | 0 | 0
  Any TEAE leading to drug interruption | 1 | 0 | 1 | 0 | 0
  Any TEAE leading to drug discontinuation | 6 | 1 | 4 | 2 | 2
  Any TEAE leading to death | 0 | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the first dose of investigational product up to 2 weeks after the end of the study (Visit 6) (approximately 6 weeks).
Description: The safety analysis set consisted of all patients who received at least 1 dose of investigational product during the study.
Arm/Group | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | RPL554 6.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/81 | 1/81 | 0/82 | 1/80 | 0/79
Serious Adverse Events (participants affected / at risk) | 2/81 | 2/81 | 1/82 | 1/80 | 1/79
Other Adverse Events (participants affected / at risk) | 20/81 | 25/81 | 24/82 | 19/80 | 25/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPL554 0.75 mg (N=81) | RPL554 1.5 mg (N=81) | RPL554 3.0 mg (N=82) | RPL554 6.0 mg (N=80) | Placebo (N=79)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPL554 0.75 mg (N=81) | RPL554 1.5 mg (N=81) | RPL554 3.0 mg (N=82) | RPL554 6.0 mg (N=80) | Placebo (N=79)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (5) | 4 (4) | 5 (5) | 7 (7)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 3 (3) | 3 (3) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 6 (6) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 5 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 7 (8) | 4 (5) | 3 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 2 (3) | 1 (1) | 4 (4) | 3 (4) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (3) | 0 (0) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator and Institution may only publish their center study activities and/or study data with prior written approval of the Sponsor.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT03443414/SAP_000.pdf
  • Study Protocol (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT03443414/Prot_001.pdf